CLINICAL TRIAL: NCT04819230
Title: Attention and Interpretation Bias Modification for Aggression Difficulties
Brief Title: A Cognitive Bias Modification RCT for Aggression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Michael McCloskey, Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27093
Record Dates: First submitted 2021-03-05; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Intermittent Explosive Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in the control condition will see the same stimuli with a different contingency for correct vs incorrect response on the computerized training task (participant masking)
  Outcome assessors will not be involved in administration of the intervention and will not be informed of participant condition (outcomes assessor masking)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bias Modification (Experimental): Attention (ATT) and interpretation (ITT) bias training. Participants complete the ATT and ITT tasks twice per week for four weeks. The ATT trains attention toward neutral stimuli and away from negative stimuli. On trials with one neutral and one threat word, the probe will always follow the location of the neutral word. Therefore, there is a contingency between the valence of the word and the location of the probe. Participants will be asked to indicate which type of probe had appeared in each trial by pressing a corresponding button as rapidly and accurately as possible. The ITT trains participants to make benign (vs. threatening) interpretations of socially-ambiguous scenarios. For each trial, a word suggesting a socially threatening or benign interpretation is presented then replaced by a sentence describing a socially-ambiguous scenario. Participants indicate if they thought the word and sentence were related. Participants will receive corrective feedback after each trial.
  Interventions: Behavioral: Cognitive Bias Modification
- Control Condition (Placebo Comparator): A combination of attention (ATT-C) and interpretation (ITT-C) control tasks
  These tasks are identical to the experimental tasks (ATT and ITT) with the exceptions that:
  ATT-C: It is designed to train attention toward neither neutral nor the threat stimuli. This will be achieved by having an equal number of probes follow the location of the threatening word and the neutral word.
  ITT-C: It is not designed to train benign interpretations of ambiguous social scenarios. Thus, no feedback will be given during the inter-trial interval, rather participants will see a blank screen between trials.
  Participants will complete both the ATT-C and ITT-C tasks twice per week for four weeks, totaling to eight experimental sessions.
  Interventions: Behavioral: Cognitive Bias Control

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — A four-week computerized attentional and interpretive bias modification protocol in which participants complete both ATT and ITT tasks twice per week, totaling to eight experimental sessions (see experimental arm for more detail.)
  Arms: Bias Modification
Behavioral: Cognitive Bias Control — A four-week computerized attentional and interpretive stimuli protocol in which participants complete both ATT-C and ITT-C tasks twice per week, totaling to eight control sessions (see placebo control arm for more detail.)
  Arms: Control Condition

SUMMARY:
This randomized controlled trial will test a computerized cognitive bias modification program (CBM) to treat attention and interpretive biases in patients with primary aggression.

DETAILED DESCRIPTION:
The objective of the proposed study is to test a computerized cognitive bias modification program (CBM) to treat attention and interpretive biases in patients with Intermittent Explosive Disorder, a disorder characterized by habitual engagement in aggressive behavior. Efficacy of the CBM program will be assessed via a small randomized controlled trial comparing CBM to a computerized control condition. This training program would consist of a four-week regimen of twice-weekly 30-minute sessions (8 sessions total) during which individuals would learn to: (a) focus attention away from threatening words toward neutral words [attention bias], and (b) to disambiguate ambiguous interpersonal scenarios using more benign, rather than threatening, interpretations [interpretive bias]. Participants will be asked to complete behavioral measures of attention bias and interpretive bias, as well as self-report measures of anger / aggression, interpretive bias, emotion regulation and life satisfaction at baseline (pre-training), post-training, and 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for current IED, as assessed via phone screen and confirmed during an in-person diagnostic interview conducted during visit one of the study
* Are able and willing to cooperate with study protocol; i.e. keep appointments, read and understand consent form, etc.
* Have written and verbal English proficiency for understanding consent and study materials

Exclusion Criteria:

* Have a lifetime history of psychosis
* Have current moderate to severe substance use disorder
* Have a history of bipolar disorder
* Have current major depressive disorder
* Are younger than 18 or older than 55 years old
* Are currently (past month) receiving treatment for anger or aggression
* Recently (past month) started or changed psychotropic medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in a Aggression from pretreatment to end of treatment (4 weeks later) and 1-month follow-up | preatment, post-treatment (4 weeks later) and 1-month follow-up. Total of 2 months
  Overt Aggression Scale-Modified (higher score means more aggression)
Change in a Anger from pretreatment to end of treatment (4 weeks later) and 1-month follow-up | pretreatment, posttreatment (4 weeks later) and 1-month follow-up. Total of 2 months
  State-Trait Anger Expression Inventory-2:state anger scale modified(higher score means more anger)
Change in Social Information Processing from pretreatment to end of treatment (4 weeks later) and 1-month follow-up | pretreatment, posttreatment (4 weeks later) and 1-month follow-up. Total of 2 months
  Social Information Processing - Attribution and Emotional Response Questionnaire

SECONDARY OUTCOMES:
Change in Emotion Regulation from pretreatment to end of treatment (4 weeks later) and 1-month follow-up | pretreatment, posttreatment (4 weeks later) and 1-month follow-up. Total of 2 months
  Difficulty in Emotion Regulation Scale (higher score means greater emotion dysregulation)
Change in IED diagnosis from pretreatment to end of treatment (4 weeks later) and 1-month follow-up | pretreatment, posttreatment (4 weeks later) and 1-month follow-up. Total of 2 months
  Intermittent Explosive Disorder-Module (presence vs absence of current disorder)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided